CLINICAL TRIAL: NCT00644111
Title: Post-operative Epidural Analgesia After Minimally Invasive Lumbar Decompression and Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHN 07-0736-A
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Low Back Pain
Keywords: Minimally Invasive Decompression and Fusion; Postoperative analgesia; Epidural; Lumbar
MeSH Terms: conditions — Low Back Pain | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Control group receiving saline placebo through an epidural catheter
  Interventions: Drug: Saline Placebo
- 2 (Active Comparator): Experimental group receiving active medication through the epidural catheter
  Interventions: Drug: Bupivicaine, Hydromorphone

INTERVENTIONS:
Drug: Bupivicaine, Hydromorphone — 0.1% Bupivicaine with 0.015mg hydromorphone per mL at 6 mL per hour in Arm 2
  Arms: 2
Drug: Saline Placebo — Saline placebo continuous epidural infusion of 6 mL per hour in Arm 1
  Arms: 1

SUMMARY:
Minimally invasive (MIS) lumbar decompression and fusion is a new procedure that aims to reduce post-operative pain, opioid consumption and related side effects, and length of hospital stay. Current research demonstrates a modest improvement in these areas beginning on the third post-operative day. MIS fusion, however, incurs significant cost as the average time of the procedure is approximately one third greater (from 148 minutes to 191 on average). Epidural analgesia has clearly demonstrated benefits for conventional open laminectomy. In order to fully maximize the benefits of an MIS technique, early post-operative analgesia/pain must be improved. The aim of this study is to combine two techniques to ultimately improve patient outcomes and satisfaction. This will be a randomized trial involving 32 patients undergoing MIS decompression and fusion with half the study group receiving active epidural and IV-PCA and the other half receiving epidural placebo and IV-PCA.

The hypothesis is that epidural analgesia will reduce post-operative opioid consumption, improve pain scores, and decrease time to ambulation as well as discharge from hospital after MIS decompression and fusion.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo minimally invasive lumbar decompression and fusion at the Toronto Western Hospital
* both genders
* ASA I to III
* BMI less than 35

Exclusion Criteria:

* refuses treatment randomization
* inability to give informed consent
* language barrier
* local anesthetic allergy
* allergy to shellfish or eggs
* bleeding diathesis
* sickle cell disease or trait
* pregnancy
* drug addiction
* psychiatric history
* severe intercurrent illness (ASA IV or V)
* patients requiring anesthesia of other surgical sites

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Reduction in opioid consumption in the first 48 hours post-operatively | 48 hours

SECONDARY OUTCOMES:
Reduction in VRS pain scores | Duration of Admission
Reduction in total opioid consumption | Duration of Admission
Reduction in opioid related side effects | Duration of Admission
Reduction in time to discharge | Duration of Admission

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD, Principal Investigator — Resident Physician, Deparment of Anesthesia, University of Toronto; Richard T Brull, MD, Principal Investigator — Department of Anesthesia, University Health Network, Toronto Western Hospital; Yoga R Rampersaud, MD, Principal Investigator — Deparment of Surgery, Division of Orthopedics, University Health Network, Toronto Western Hospital; Vincent WS Chan, MD, Study Director — Department of Anesthesia, University Health Network, Toronto Western Hospital; Paul S Tumber, MD, Study Director — Department of Anesthesia, University Health Network, Toronto Western Hospital
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kundra P, Gurnani A, Bhattacharya A. Preemptive epidural morphine for postoperative pain relief after lumbar laminectomy. Anesth Analg. 1997 Jul;85(1):135-8. doi: 10.1097/00000539-199707000-00024. PMID 9212136
- [Background] Schenk MR, Putzier M, Kugler B, Tohtz S, Voigt K, Schink T, Kox WJ, Spies C, Volk T. Postoperative analgesia after major spine surgery: patient-controlled epidural analgesia versus patient-controlled intravenous analgesia. Anesth Analg. 2006 Nov;103(5):1311-7. doi: 10.1213/01.ane/0000247966.49492.72. PMID 17056975
- [Background] Turner A, Lee J, Mitchell R, Berman J, Edge G, Fennelly M. The efficacy of surgically placed epidural catheters for analgesia after posterior spinal surgery. Anaesthesia. 2000 Apr;55(4):370-3. doi: 10.1046/j.1365-2044.2000.01117.x. PMID 10781125
- [Background] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Background] Gottschalk A, Freitag M, Tank S, Burmeister MA, Kreil S, Kothe R, Hansen-Algenstedt N, Weisner L, Staude HJ, Standl T. Quality of postoperative pain using an intraoperatively placed epidural catheter after major lumbar spinal surgery. Anesthesiology. 2004 Jul;101(1):175-80. doi: 10.1097/00000542-200407000-00027. PMID 15220788
- [Background] Blumenthal S, Min K, Nadig M, Borgeat A. Double epidural catheter with ropivacaine versus intravenous morphine: a comparison for postoperative analgesia after scoliosis correction surgery. Anesthesiology. 2005 Jan;102(1):175-80. doi: 10.1097/00000542-200501000-00026. PMID 15618801
- [Background] Ray CD, Bagley R. Indwelling epidural morphine for control of post-lumbar spinal surgery pain. Neurosurgery. 1983 Oct;13(4):388-93. doi: 10.1227/00006123-198310000-00007. PMID 6633831
- [Background] Cohen BE, Hartman MB, Wade JT, Miller JS, Gilbert R, Chapman TM. Postoperative pain control after lumbar spine fusion. Patient-controlled analgesia versus continuous epidural analgesia. Spine (Phila Pa 1976). 1997 Aug 15;22(16):1892-6; discussion 1896-7. doi: 10.1097/00007632-199708150-00016. PMID 9280026
- [Background] Fisher CG, Belanger L, Gofton EG, Umedaly HS, Noonan VK, Abramson C, Wing PC, Brown J, Dvorak MF. Prospective randomized clinical trial comparing patient-controlled intravenous analgesia with patient-controlled epidural analgesia after lumbar spinal fusion. Spine (Phila Pa 1976). 2003 Apr 15;28(8):739-43. PMID 12698113
- [Background] Park Y, Ha JW. Comparison of one-level posterior lumbar interbody fusion performed with a minimally invasive approach or a traditional open approach. Spine (Phila Pa 1976). 2007 Mar 1;32(5):537-43. doi: 10.1097/01.brs.0000256473.49791.f4. PMID 17334287
- [Background] Podichetty VK, Spears J, Isaacs RE, Booher J, Biscup RS. Complications associated with minimally invasive decompression for lumbar spinal stenosis. J Spinal Disord Tech. 2006 May;19(3):161-6. doi: 10.1097/01.bsd.0000188663.46391.73. PMID 16770211
- [Background] Sandhu NS, Sidhu DS, Capan LM. The cost comparison of infraclavicular brachial plexus block by nerve stimulator and ultrasound guidance. Anesth Analg. 2004 Jan;98(1):267-268. doi: 10.1213/01.ANE.0000077685.55641.7C. No abstract available. PMID 14693638
- [Background] Brull R, McCartney CJ, Chan VW, El-Beheiry H. Neurological complications after regional anesthesia: contemporary estimates of risk. Anesth Analg. 2007 Apr;104(4):965-74. doi: 10.1213/01.ane.0000258740.17193.ec. PMID 17377115
- [Background] Foley KM. The treatment of cancer pain. N Engl J Med. 1985 Jul 11;313(2):84-95. doi: 10.1056/NEJM198507113130205. PMID 2582259
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Derived] Choi S, Rampersaud YR, Chan VW, Persaud O, Koshkin A, Tumber P, Brull R. The addition of epidural local anesthetic to systemic multimodal analgesia following lumbar spinal fusion: a randomized controlled trial. Can J Anaesth. 2014 Apr;61(4):330-9. doi: 10.1007/s12630-014-0115-z. Epub 2014 Feb 12. PMID 24519631